CLINICAL TRIAL: NCT04585737
Title: Efficacy, Safety and Tolerability of Switching to Dolutegravir/Lamivudine in Virologically-suppressed Adults Living With HIV on Bictegravir/Tenofovir Alafenamide/emtricitabine-the DYAD Study
Brief Title: Efficacy of Switching to DTG/3TC in Virologically-suppressed Adults Currently on B/F/TAF
Acronym: DYAD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charlotte-Paige Rolle, MD (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor-Investigator, Charlotte-Paige Rolle, MD, Principal Investigator, Orlando Immunology Center
Organization: Orlando Immunology Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OIC 008
Record Dates: First submitted 2020-09-22; First posted 2020-10-14 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-09

CONDITIONS: HIV I Infection
Keywords: switch study; dovato; biktarvy
MeSH Terms: interventions — dolutegravir; Lamivudine; bictegravir; Emtricitabine; tenofovir alafenamide; bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Intervention Model Description: Randomized, open-label, active-controlled study of virologically suppressed participants living with HIV
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment group 1 (Experimental): Treatment Group 1 (n=148): FDC of DTG/3TC (50mg/300mg) administered orally, once daily (QD), without regard to food.
  Interventions: Drug: Dolutegravir / Lamivudine Pill
- Treatment group 2 (Active Comparator): Treatment Group 2 (n=74): Stay on baseline regimen consisting of FDC of B/F/TAF (50mg/200mg/ 25mg) (taken as prescribed) without regard to food.
  Interventions: Drug: Bictegravir / Emtricitabine / Tenofovir Alafenamide Pill

INTERVENTIONS:
Drug: Dolutegravir / Lamivudine Pill — Experimental
  Other Names: Dovato
  Arms: Treatment group 1
Drug: Bictegravir / Emtricitabine / Tenofovir Alafenamide Pill — Active comparator
  Other Names: Biktarvy
  Arms: Treatment group 2

SUMMARY:
Phase 4, randomized, open-label study to evaluate the efficacy, safety and tolerability of switching virologically suppressed adults living with HIV on bictegravir/tenofovir alafenamide/emtricitabine to dolutegravir/lamivudine

DETAILED DESCRIPTION:
Randomized, open-label, active-controlled study of virologically suppressed participants living with HIV

Participants who provide written informed consent and meet all the eligibility criteria will be randomized in a 2:1 ratio to one of the following 2 treatment groups:

Treatment Group 1 (n=148): FDC of DTG/3TC (50mg/300mg) administered orally, once daily (QD), without regard to food.

Treatment Group 2 (n=74): Stay on baseline regimen consisting of FDC of B/F/TAF (50mg/200mg/ 25mg) (taken as prescribed) without regard to food.

Randomization will be stratified by gender and race at entry given that this study aims to enroll at least 30% of participants who are female and African American.

All participants will be responsible for using their insurance plan to obtain coverage for DTG/3TC and or B/F/TAF, in addition to any labs required by the study. This expectation is clearly outlined in the informed consent. The study team will work with participants to minimize their co-pays for study medications and labs through the use of manufacturer and other external assistance programs.

Study duration will be 48 weeks.

Number of participants planned: Approximately 222 participants

Target Population: HIV-1 infected adult participants who are virologically suppressed (HIV-1 RNA<50 copies/mL) on FDC of B/F/TAF (50mg/200mg/ 25mg) ≥ 3 months prior to screening

ELIGIBILITY:
Inclusion Criteria -

1. Aged 18 years or older at the time of signing the informed consent

   TYPE OF SUBJECT AND DIAGNOSIS INCLUDING DISEASE SEVERITY
2. HIV-1 infected men or women.
3. Must have a stable form of insurance that is expected to continue without significant changes for at least 48 weeks
4. Documented evidence of at least two plasma HIV-1 RNA measurements <50 c/mL at least 3 months apart prior to Day 1 (the screening HIV-1 RNA can count as the second measurement)
5. Plasma HIV-1 RNA <50 c/mL at Screening.
6. Must be on uninterrupted B/F/TAF for at least 3 months prior to screening

   SEX
7. Male or female A female subject is eligible to participate if she is not pregnant [as confirmed by a negative serum human chorionic gonadotrophin (hCG) test at screen and a negative urine hCG test at Day

1/Randomization (a local serum hCG test at Randomization is allowed if it can be done, and results obtained, within 24 hours prior to randomization)], not lactating, and at least one of the following conditions applies:

1. Non-reproductive potential defined as:

   * Pre-menopausal females with one of the following:

     o Documented tubal ligation
     * Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion
     * Hysterectomy
     * Documented Bilateral Oophorectomy
   * Post-menopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause (refer to laboratory reference ranges for confirmatory levels)]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study.

   Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment.
2. Reproductive potential and agrees to follow one of the options listed in the Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) (see Appendix 2) from 30 days prior to the first dose of study medication and for at least 2 weeks after the last dose of study medication.

The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception. All subjects participating in the study should be counseled on safer sexual practices including the use and benefit/risk of effective barrier methods (e.g., male condom) and on the risk of HIV transmission to an uninfected partner.

INFORMED CONSENT

8. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the consent form and in this protocol. Eligible subjects must sign a written Informed Consent Form before any protocol-specified assessments are conducted

b. Exclusion Criteria

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

Exclusion Criteria -

CONCURRENT CONDITIONS/MEDICAL HISTORY

1. Women who are breastfeeding or plan to become pregnant or breastfeed during the study.
2. Any evidence of an active Centers for Disease Control and Prevention (CDC) Stage 3 disease [15], EXCEPT cutaneous Kaposi's sarcoma not requiring systemic therapy. Historical or current CD4 cell counts less than 200 cells/mm3 are NOT exclusionary.
3. Subjects with severe hepatic impairment (Class C) as determined by Child-Pugh classification [16].
4. Unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, esophageal or gastric varices, or persistent jaundice), cirrhosis, known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
5. Evidence of Hepatitis B virus (HBV) infection based on the results of testing at Screening for Hepatitis B surface antigen (HBsAg), Hepatitis B core antibody (antiHBc), Hepatitis B surface antigen antibody (anti-HBs) and HBV DNA as follows:

   * Subjects positive for HBsAg are excluded.
   * Subjects negative for anti-HBs but positive for anti-HBc (negative HBsAg status) and positive for HBV DNA are excluded.

   Note: Subjects positive for anti-HBc (negative HBsAg status) and positive for antiHBs (past and/or current evidence) are immune to HBV and are not excluded. AntiHBc must be either total anti-HBc or anti-HBc immunoglobulin G (IgG), and NOT anti-HBc IgM.
6. Anticipated need for any hepatitis C virus (HCV) therapy during the first 48 weeks of the study
7. Untreated syphilis infection (positive rapid plasma reagin [RPR] at Screening without clear documentation of treatment). Subjects who are at least 7 days post completed treatment are eligible.
8. History or presence of allergy or intolerance to the study drugs or their components or drugs of their class.
9. Ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous cell carcinoma, or cervical, anal or penile intraepithelial neoplasia.
10. Subjects who in the investigator's judgment, poses a significant suicidality risk.

    EXCLUSIONARY TREATMENTS PRIOR TO SCREENING OR DAY 1
11. Treatment with an HIV-1 immunotherapeutic vaccine within 90 days of Screening
12. Treatment with any of the following agents within 28 days of Screening

    * radiation therapy
    * cytotoxic chemotherapeutic agents
    * any systemic immune suppressant
13. Exposure to an experimental drug or experimental vaccine within either 28 days, 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent, whichever is longer, prior to the first dose of study medication.
14. Use of any regimen consisting of single or dual ART LABORATORY VALUES OR CLINICAL ASSESSMENTS AT SCREENING
15. Any evidence of major NRTI mutation (defined as history of 3 or more TAMs (M41L, D67N, K70R, L210W, T215F/Y, and K219Q/E/N/R), M184V/I, T69-insertions, or K65R/E/N) or presence of any major INSTI resistance-associated mutation [17] in any available prior resistance genotype assay test result
16. Any verified Grade 4 laboratory abnormality
17. Alanine aminotransferase (ALT) ≥5 times the upper limit of normal (ULN) or ALT ≥3xULN and bilirubin ≥1.5xULN (with >35% direct bilirubin).
18. Creatinine clearance of <50mL/min/1.73m2 via CKD-EPI method.

    EXCLUSIONARY CRITERIA PRIOR TO SCREENING OR DAY 1
19. Within the 6 to 12-month window prior to Screening and after confirmed suppression to <50 copies/mL, any plasma HIV-1 RNA measurement >200 c/mL.
20. Within the 6 to 12-month window prior to Screening and after confirmed suppression to <50 copies/mL, 2 or more plasma HIV-1 RNA measurements ≥50 c/mL.
21. Within 6 months prior to Screening and after confirmed suppression to <50 c/mL on current ART regimen, any plasma HIV-1 RNA measurement ≥50 copies/mL.
22. Any drug holiday during the 12 months prior to Screening, except for brief periods (less than 1 month) where all ART was stopped due to tolerability and/or safety concerns.
23. Any history of switch to another regimen, defined as change of a single drug or multiple drugs simultaneously, due to virologic failure to therapy (defined as a confirmed plasma HIV-1 RNA ≥400 copies/mL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte-Paige Rolle, MD, Principal Investigator — Orlando Immunology Center
Locations (1):
- Orlando Immunology Center, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant was screened on 10/5/2020 and the last participant's Week 48 visit was on 8/3/2023. Of 235 screened, 222 were enrolled and randomized to switch to DTG/3TC (n=149) or continue B/F/TAF (n=73), 222 received study treatment (ITT-E)
Groups:
- Treatment Group 1: Treatment Group 1 (n=149): FDC of DTG/3TC (50mg/300mg) administered orally, once daily (QD), without regard to food.
  Dolutegravir / Lamivudine Pill: Experimental
- Treatment Group 2: Treatment Group 2 (n=73): Stay on baseline regimen consisting of FDC of B/F/TAF (50mg/200mg/ 25mg) (taken as prescribed) without regard to food.
  Bictegravir / Emtricitabine / Tenofovir Alafenamide Pill: Active comparator
Period: Overall Study
Arm/Group | Treatment Group 1 | Treatment Group 2
Started | 149 | 73
Completed | 133 | 65
Not Completed | 16 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group 1 | Treatment Group 2 | Total
Number analyzed (Participants) | 149 | 73 | 222
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 140 | 62 | 202
  >=65 years | 9 | 11 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 12 | 36
  Male | 125 | 61 | 186
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 102 | 54 | 156
  Black/African American | 44 | 18 | 62
  Other | 3 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 149 | 73 | 222

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Measure is to Evaluate the Efficacy of Switching From B/F/TAF to DTG/3TC Versus Continuing B/F/TAF as Determined by the Proportion of Participants With HIV-1 RNA ≥50 Copies/mL at Week 48
Description: percentage with HIV-1 RNA ≥50 copies/mL at Week 48 in each treatment arm
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group 1 | Treatment Group 2
Number analyzed (Participants) | 149 | 73
Participants | 6 | 5

2. Secondary Outcome: The Secondary Outcome Measure is to Evaluate the Efficacy of Switching to DTG/3TC From B/F/TAF as Determined by the Proportion of Participants With HIV-1 RNA≥ 50 Copies/mL at Week 24
Description: percentage with HIV-1 RNA ≥50 copies/mL at Week 24 in each treatment arm
Time Frame: 24 weeks
Population: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group 1 | Treatment Group 2
Number analyzed (Participants) | 149 | 73
Participants | 3 | 3

3. Secondary Outcome: The Secondary Outcome Measure is to Evaluate the Efficacy of Switching to DTG/3TC From B/F/TAF as Determined by the Proportion of Participants With HIV-1 RNA<50 Copies/mL at Week 48
Description: percentage with HIV-1 RNA<50 copies/mL at Weeks 12, 24 and 48 in each treatment arm
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group 1 | Treatment Group 2
Number analyzed (Participants) | 149 | 73
Participants | 127 | 59

4. Secondary Outcome: The Secondary Outcome Measure is to Measure the Incidence and Severity of Grade 2-5 Drug-related Adverse Events and Laboratory Abnormalities (Graded Using DAIDs Grading Scale) Through 48 Weeks
Description: Grade 2-5 drug-related AEs and lab abnormalities graded using DAIDS grading scale
Time Frame: 48 weeks
Population: overall number of participants experiencing Grade 2-5, drug-related AEs
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group 1 | Treatment Group 2
Number analyzed (Participants) | 149 | 73
Participants | 14 | 1

5. Secondary Outcome: The Secondary Outcome Measure is to Evaluate the Proportion of Participants That Discontinue Treatment Through 48 Weeks in Each Treatment Arm and Reasons for Discontinuation
Description: Number of participants who discontinue study treatment and reasons for discontinuation
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group 1 | Treatment Group 2
Number analyzed (Participants) | 149 | 73
Participants | 15 | 9

6. Secondary Outcome: The Secondary Outcome Measure is to Evaluate the Effects of DTG/3TC Once Daily on Fasting Total Cholesterol Over Time Compared to B/F/TAF Through 48 Weeks
Description: Change from Baseline in fasting total cholesterol at Week 48
Time Frame: 48 weeks
Population: change in total cholesterol
Measure: Mean (Full Range); unit: mg/dL
Arm/Group | Treatment Group 1 | Treatment Group 2
Number analyzed (Participants) | 149 | 73
mg/dL | -2.3 [-11.5 to 21.3] | 3.3 [-19 to 33.5]

7. Secondary Outcome: The Secondary Outcome Measure is to Evaluate Changes in Weight (kg) in Those Treated With DTG/3TC vs. B/F/TAF Over Time
Description: Change from Baseline in weight (kg) measured at Week 48
Time Frame: 48 weeks
Population: mean change in weight at 48 weeks
Measure: Mean (Full Range); unit: kg
Arm/Group | Treatment Group 1 | Treatment Group 2
Number analyzed (Participants) | 149 | 73
kg | -1 [-7.3 to 4.3] | 0.2 [-5.8 to 6.1]

8. Secondary Outcome: The Secondary Outcome Measure is to Evaluate Changes in Waist Circumference (Inches) in Those Treated With DTG/3TC vs. B/F/TAF Over Time
Description: Change from Baseline in waist circumference (measured in inches) at Week 48
Time Frame: 48 weeks
Population: mean change from baseline in weight circumference
Measure: Mean (Full Range); unit: inches
Arm/Group | Treatment Group 1 | Treatment Group 2
Number analyzed (Participants) | 149 | 73
inches | -0.9 [-1.6 to 2.3] | -0.7 [-2.1 to 3.8]

9. Secondary Outcome: The Secondary Outcome Measure is to Evaluate Changes in BMI (kg/m2) in Those Treated With DTG/3TC vs. B/F/TAF Over Time
Description: Change from Baseline in weight (kg) and height (meters) will be used to assess changes in BMI (kg/m2) measured at Week 48
Time Frame: 48 weeks
Population: change in BMI over 48 weeks
Measure: Mean (Full Range); unit: kg/m2
Arm/Group | Treatment Group 1 | Treatment Group 2
Number analyzed (Participants) | 149 | 73
kg/m2 | -0.6 [-1.1 to 0.9] | -0.1 [-1.3 to 1.6]

10. Secondary Outcome: To Assess the Number of Subjects With Genotypic Mutations Affecting Any Component of the Treatment Regimen Among Subjects Meeting Virologic Rebound Criteria (HIV-1 RNA≥50 Copies/mL X2) Using HIV Genotypic and ARCHIVE HIV-DNA Testing
Description: to measure the incidence of observed genotypic resistance to ARVs for subjects meeting Virologic Rebound Criteria
Time Frame: 48 weeks
Population: number of participants with treatment-emergent resistance through Week 48
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group 1 | Treatment Group 2
Number analyzed (Participants) | 12 | 6
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: 48 weeks
Description: Additional secondary endpoints included safety and tolerability which were evaluated through incidence and severity of AEs, laboratory abnormalities and discontinuations due to AEs at each study visit through Week 48.
Arm/Group | Treatment Group 1 | Treatment Group 2
All-Cause Mortality (participants affected / at risk) | 0/149 | 0/73
Serious Adverse Events (participants affected / at risk) | 12/149 | 4/73
Other Adverse Events (participants affected / at risk) | 14/149 | 1/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group 1 (N=149) | Treatment Group 2 (N=73)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) — This was the only drug-related SAE and occurred in the DTG/3TC arm
COVID-19 (Infections and infestations) | 0 | 3
Chest Pain (Cardiac disorders) | 2 | 1
Drug Overdose (Psychiatric disorders) | 1 | 0
Bipolar Disorder (Psychiatric disorders) | 1 | 0
Left hip pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cellulitis (Infections and infestations) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Fall (Musculoskeletal and connective tissue disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group 1 (N=149) | Treatment Group 2 (N=73)
Nausea (Gastrointestinal disorders) | 7 | 0 — Drug related, Grade 2-5
Fatigue (General disorders) | 6 | 0 — Drug-related, Grade 2-5
Diarrhea (Gastrointestinal disorders) | 5 | 0 — Drug-related, Grade 2-5
Headaches (Nervous system disorders) | 5 | 0 — Drug-related, grade 2-5
Insomnia (Nervous system disorders) | 5 | 0 — Drug-related, Grade 2-5
Worsening depression (Psychiatric disorders) | 3 | 0 — Drug-related, Grade 2-5
Dizziness (Nervous system disorders) | 3 | 0 — Drug-related, Grade 2-5
Constipation (Gastrointestinal disorders) | 2 | 1 — Drug-related, Grade 2-5
Proteinuria (Renal and urinary disorders) | 0 | 1 — Drug-related, Grade 2-5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-29): https://cdn.clinicaltrials.gov/large-docs/37/NCT04585737/Prot_SAP_000.pdf